CLINICAL TRIAL: NCT03940781
Title: Effects of Rehabilitation for Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hsia Hung, Department chairman of physical therapy, College of Medicine, National Cheng Kung University, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKUH-10802018
Record Dates: First submitted 2019-01-10; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: obstructive sleep apnea; oropharyngeal rehabilitation; cardiopulmonary rehabilitation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: 30 participants with moderate or severe OSA (AHI≥15) were randomized into intervention group (N=15) and control group (N=15).
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and assessors blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): We conducted a twice a week, 12-week-intervention of 'comprehensive rehabilitation'
  Interventions: Behavioral: comprehensive rehabilitation
- control group (No Intervention): We kept the patients for the waiting list until after completing baseline and 12-week measurement

INTERVENTIONS:
Behavioral: comprehensive rehabilitation — oropharyngeal rehabilitation, cardiopulmonary rehabilitation, and therapeutic exercise
  Arms: intervention group

SUMMARY:
In previous review study, it was hypothesized that a comprehensive rehabilitation can combine both local pharyngeal muscle exercise and systemic cardiopulmonary rehabilitation for the OSA patients with oropharyngeal muscle dysfunction or ventilator drive instability. To develop a comprehensive rehabilitation model is of innovative care strategy in this study.

DETAILED DESCRIPTION:
BACKGROUND: Obstructive sleep apnea (OSA) is a prevalent sleep-related breathing disorder, which was characterized by repetitive events of complete and partial obstructions of the upper airway. The pathogenesis of OSA is interacted by multiple factors, primarily including upper airway (UA) anatomic impairment, ventilatory drive instability, and oropharyngeal muscle dysfunction. However, studies have proven prior oropharyngeal exercise was designed for those OSA patients with oropharyngeal muscle dysfunction. Unlike prior oropharyngeal exercise, comprehensive rehabilitation should emphasize the cardiorespiratory regulation capability in addition to oropharyngeal function.

OBJECTIVES: Therefore, the purpose of this study is to explore both the clinical and biological effects of our comprehensive rehabilitation, we used PSG data as clinical effect and biomarker of inflammation expression as biological effect.

METHODS: Thirty subjects with moderate or severe OSA (AHI≥15) were randomized into intervention group (N=15) and control group (N=15). In intervention group, a 12-week-intervention of out-patient rehabilitation program included oropharyngeal muscle training, threshold respiratory muscle training, and therapeutic exercise.

ANTICIPATED OUTCOMES: The preliminary results would demonstrate promisingly clinical effects and biological effects of our comprehensive rehabilitation model. Therefore, the further studies should emphasize the methods to differentiate diagnosis for the indicated patients with oropharyngeal muscle dysfunction or ventilatory drive instability.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35-65 with or without surgery had difficulty accepting or adhering CPAP

Exclusion Criteria:

* BMI<32
* Smoking or alcoholism
* Severe allergic rhinitis
* Stroke history
* CVD
* Severe restricted or obstructive pulmonary disease
* Hypothyroidism
* DM or HTN without stable control
* Psychiatric disease
* Co-existing non-respiratory sleep disorders

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopea-index | Change from Baseline Apnea-hypopnea-index at 12 weeks
  average apnea and hypopnea events per hour during sleep test
potential biomarkers of endothelial dysfunction | at 12 weeks
  count of ICAM-1, VCAM-1, and NF-κB molecule in plasma serum (%)

SECONDARY OUTCOMES:
Oropharyngeal muscle function | at 12 weeks
  myofunctional scale of genioglossus muscles, mastication muscles, and deglultition muscles
Respiratory muscle function | at 12 weeks
  PImax(mmH2O), PEmax(mmH2O)
Respiratory muscle function | at 12 weeks
  pulmonary function test (FVC%,FEV1%,FEF50%,FIF50%)
Hear rate variability | at 12 weeks
  time domain and frequency domain HRV

CONTACTS AND LOCATIONS:
Overall Officials: Chinghsia Hung, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No